CLINICAL TRIAL: NCT00427960
Title: A Phase IV, 6-week, Randomised, Double-blind, Multicentre, Parallel Group, Comparative Study to Evaluate the Efficacy of Rosuvastatin 5mg and Atorvastatin 10mg in UK Asian Subjects With Primary Hypercholesterolaemia
Brief Title: Study of Asian Patients With Hypercholesterolaemia in the UK - Rosuvastatin 5mg Versus Atorvastatin 10mg
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to inadequate recruitment
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3560L00060; SHUKRA
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Results first posted 2010-03-22 (Estimated); Last update posted 2010-12-16 (Estimated); Status verified 2010-11

CONDITIONS: Hypercholesterolaemia
Keywords: cholesterol; statin; Asian; LDL-cholesterol
MeSH Terms: conditions — Hypercholesterolemia | interventions — Nutrition Assessment; Rosuvastatin Calcium; Atorvastatin

ARMS (2):
- rosuvastatin (Active Comparator): rosuvastatin 5 mg
  Interventions: Behavioral: Dietary advice; Drug: rosuvastatin
- atorvastatin (Active Comparator): atorvastatin 10 mg
  Interventions: Behavioral: Dietary advice; Drug: atorvastatin

INTERVENTIONS:
Behavioral: Dietary advice
Drug: rosuvastatin — rosuvastatin 5 mg
  Other Names: Crestor
  Arms: rosuvastatin
Drug: atorvastatin — atorvastatin 10 mg
  Arms: atorvastatin

SUMMARY:
The purpose of this study is to compare the effectiveness and safety of rosuvastatin 5mg in lowering blood cholesterol, compared to one other medicine, atorvastatin 10mg in Asian patients in the UK.

ELIGIBILITY:
Inclusion Criteria:

* Self described Asian, first or second generation
* Male or female > or = 18 years with primary hypercholesterolaemia.

Exclusion Criteria:

* Use of cholesterol lowering drugs from visit 1
* Homozygous familial hypercholesterolaemia
* Active arterial disease within 3 months of study entry
* Poorly controlled diabetes
* Uncontrolled hypothyroidism
* Active liver disease
* History of alcoh/drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rhiannon Rowsell, MD, Study Director — AstraZeneca; Shahid Ali, MD, Principal Investigator — Bradford PCT
Locations (9):
- United Kingdom (9):
  - Research Site, Allerton
  - Research Site, Birmingham
  - Research Site, Blackburn
  - Research Site, Bolton
  - Research Site, Crawley
  - Research SIte, Glasgow
  - Research Site, Newcastle
  - Research SIte, Sheffield
  - Research SIte, Slough

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 25 primary and secondary care centres in the United Kingdom. The first participant was enrolled on 20th December 2006 and the last participant entered the study on 16th November 2007.
Pre-assignment Details: Participants entered an initial 6-week dietary run-in/ wash-out period, after which those with a fasting low density lipoprotein cholesterol (LDL-C) of greater than or equal to 4.00 mmol/L and triglycerides (TG) less than 4.52 mmol/L, were randomised to receive treatment with either rosuvastatin 5 mg plus atorvatstatin , or atorvastatin 10mg
Period: Overall Study
Arm/Group | Rosuvastatin | Atorvastatin
Started | 30 | 25
Completed | 28 | 21
Not Completed | 2 | 4
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rosuvastatin | Atorvastatin | Total
Number analyzed (Participants) | 30 | 25 | 55
Age Continuous [Mean (Standard Deviation); unit: years] | 50 (11) | 53 (11) | 51.5 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24.0
  Male | 17 | 14 | 31.0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Low Density Lipoprotein - Cholesterol (LDL-C)
Description: Calculated as LDL-C at Week 6 - LDL-C at Week 12] * 100
Time Frame: 6 weeks (baseline) and 12 weeks
Population: Intention to treat (ITT) population (all randomized patients).
Measure: Number; unit: Percent Change in LDL-C
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 30 | 25
Percent Change in LDL-C | 33.28 | 36.92

2. Secondary Outcome: The Percentage of Participants Reaching the General Medical Services (GMS) Contract Target of Total Cholesterol (TC) <5 mmol/L
Time Frame: 6 weeks (Baseline) and 12 weeks
Population: Intention to treat (ITT) population (all randomized patients).
Measure: Number; unit: Percentage of Participants
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 30 | 25
Percentage of Participants | 50 | 64

3. Secondary Outcome: The Percentage of Participants Reaching the Joint British Societies' Guideline (JBS 2) Targets of TC <4 mmol/L and LDL-C <2 mmol/L
Time Frame: 6 weeks (baseline) and 12 weeks
Population: Intention to treat (ITT) population (all randomized patients).
Measure: Number; unit: Percentage of Participants
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 30 | 25
Percentage of Participants | 16 | 28

4. Secondary Outcome: The Percentage of Participants Reaching the European (EAS) Targets of LDL-C<2.5 or 3.00 mmol/L, Depending on Risk Category, and the Combined LDL-C and TC Target of LDL-C<2.5 or 3.0 mmol/L and TC<4.5 or 5.0 mmol/L, Both Depending on Risk Category.
Description: Risk categories are:
  Symptomatic Asymptomatic, total risk <5% Asymptomatic, total risk ≥5%, baseline LDL-C<3 mmol/L and baseline TC<5 mmol/L Asymptomatic, total risk ≥5%, baseline LDL-C ≥3 mmol/L or baseline TC ≥5 mmol/L
  Patients are defined as symptomatic if they meet at least 1 of the following criteria:
  History of cardiovascular disease Type II diabetes or diabetes of unknown type Baseline TC ≥8 mmol/l Baseline LDL-C ≥6 mmol/l Baseline systolic BP ≥180 mmHg Baseline diastolic BP ≥110 mmHg
  Total risk is derived from age, sex, TC, systolic BP and smoking status.
Time Frame: 6 weeks (baseline) and 12 weeks
Population: Intention to treat (ITT) population (all randomized patients).
Measure: Number; unit: Percentage of Participants
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 30 | 25
Percentage of Participants | 43 | 48

5. Secondary Outcome: The Percentage Change From Baseline(week6) in TC
Description: Derived according to the following formula: 100*[Lipid at week 12 - Lipid at week 6]/Lipid at week 6
Time Frame: 6 weeks (baseline) and 12 weeks
Population: Intention to treat (ITT) population (all randomized patients).
Measure: Number; unit: Percent Change in TC
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 30 | 25
Percent Change in TC | -23.03 | -26.88

6. Secondary Outcome: The Percentage Change From Baseline (Week 6) in High-density Lipoprotein Cholesterol (HDL-C)
Description: Derived according to the following formula: 100*[Lipid at week 12 - Lipid at week 6]/Lipid at week 6
Time Frame: 6 weeks (baseline) and 12 weeks
Population: Intention to treat (ITT) population (all randomized patients).
Measure: Number; unit: Percent Change in HDL-C
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 30 | 25
Percent Change in HDL-C | 4.46 | 3.15

7. Secondary Outcome: The Percentage of Participants Reaching the Joint British Societies Guideline (JBS 2) Target of TC <4 mmol/L
Time Frame: 6 weeks (baseline) and 12 weeks
Population: Intention to treat (ITT) population (all randomized patients).
Measure: Number; unit: Percentage of Participants
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 30 | 25
Percentage of Participants | 13 | 12

8. Secondary Outcome: The Percentage Change From Baseline (Week 6)in Non-HDL-C
Description: Derived according to the following formula: 100*[Lipid at week 12 - Lipid at week 6]/Lipid at week 6
Time Frame: 6 weeks (baseline) and 12 weeks
Population: Intention to treat (ITT) population (all randomized patients).
Measure: Number; unit: Percent Change in Non-HDL-C
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 30 | 25
Percent Change in Non-HDL-C | -29.72 | -34.09

9. Secondary Outcome: The Percentage Change From Baseline (Week 6) in Apolipoprotein-B (ApoB)
Description: Derived according to the following formula: 100*[Lipid at week 12 - Lipid at week 6]/Lipid at week 6
Time Frame: 6 weeks (baseline) and 12 weeks
Population: Intention to treat (ITT) population (all randomized patients).
Measure: Number; unit: Percent Change in ApoB
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 30 | 25
Percent Change in ApoB | -25.96 | -28.67

10. Secondary Outcome: The Percentage Change From Baseline (Week 6) in Apolipoprotein-A1 (ApoA1)
Description: Derived according to the following formula: 100*[Lipid at week 12 - Lipid at week 6]/Lipid at week 6
Time Frame: 6 weeks (baseline) and 12 weeks
Population: Intention to treat (ITT) population (all randomized patients).
Measure: Number; unit: Percent Change in ApoA1
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 30 | 25
Percent Change in ApoA1 | -0.55 | 1.89

11. Secondary Outcome: The Percentage Change From Baseline (Week 6)in LDL-C/HDL-C Ratio
Description: Derived according to the following formula: 100*[Lipid at week 12 - Lipid at week 6]/Lipid at week 6
Time Frame: 6 weeks (baseline) and 12 weeks
Population: Intention to treat (ITT) population (all randomized patients).
Measure: Number; unit: Percent Change in LDL-C/HDL-C Ratio
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 30 | 25
Percent Change in LDL-C/HDL-C Ratio | -34.75 | -38.45

12. Secondary Outcome: The Percentage Change From Baseline (Week 6) in TC/HDL-C Ratio
Description: Derived according to the following formula: 100*[Lipid at week 12 - Lipid at week 6]/Lipid at week 6
Time Frame: 6 weeks (baseline) and 12 weeks
Population: Intention to treat (ITT) population (all randomized patients).
Measure: Number; unit: Percent Change in TC/HDL-C Ratio
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 30 | 25
Percent Change in TC/HDL-C Ratio | -24.99 | -28.42

13. Secondary Outcome: The Percentage Change From Baseline(Week 6) in Non-HDL-C/HDL-C Ratio
Description: Derived according to the following formula: 100*[Lipid at week 12 - Lipid at week 6]/Lipid at week 6
Time Frame: 6 weeks (baseline) and 12 weeks
Population: Intention to treat (ITT) population (all randomized patients).
Measure: Number; unit: Percent Change in Non-HDL-C/HDL-C Ratio
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 30 | 25
Percent Change in Non-HDL-C/HDL-C Ratio | -31.05 | -35.48

14. Secondary Outcome: The Percentage Change From Baseline (Week 6) in ApoB/ApoA1 Ratio
Description: Derived according to the following formula: 100*[Lipid at week 12 - Lipid at week 6]/Lipid at week 6
Time Frame: 6 weeks (baseline) and 12 weeks
Population: Intention to treat (ITT) population (all randomized patients).
Measure: Number; unit: Percent Change in ApoB/ApoA1 Ratio
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 30 | 25
Percent Change in ApoB/ApoA1 Ratio | -22.89 | -28.75

15. Secondary Outcome: The Percentage of Participants Reaching the European (EAS) Targets of LDL-C<2.5 or 3.00 mmol/L, Depending on Risk Category.
Description: as for outcome 4
Time Frame: 6 weeks (baseline) and 12 weeks
Population: Intention to treat (ITT) population (all randomized patients).
Measure: Number; unit: Percentage of Participants
Arm/Group | Rosuvastatin | Atorvastatin
Number analyzed (Participants) | 30 | 25
Percentage of Participants | 56.7 | 56.0

ADVERSE EVENTS:
Arm/Group | Rosuvastatin | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 1 | 0
Other Adverse Events (participants affected / at risk) | 4 | 3
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Rosuvastatin | Atorvastatin
Cerebrovascular Accident (Nervous system disorders) | 1/30 | 0/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Rosuvastatin | Atorvastatin
Dizziness (Nervous system disorders) | 3/30 | 1/25
Headache (Nervous system disorders) | 1/30 | 2/25

LIMITATIONS AND CAVEATS:
The study achieved only 8% of the randomised target number of patients and for this reason alone was terminated early. Planned statistical analyses could not be performed. No scientifically valid conclusions can be drawn from the limited study data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other